CLINICAL TRIAL: NCT06656832
Title: Peripheral Drivers of Heart Failure Progression - the Prospective PEDAL-HF Study
Acronym: PEDAL-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 242/24-ek; 934700-034 (Other: Universität Leipzig)
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure - NYHA II - IV
Keywords: Heart Failure Network Care

STUDY DESIGN:
Masking Description: The primary endpoint (NT-proBNP) will be measured by lab personnel blinded to patients´ group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Randomised Arm 1: Heart Failure Network Care (Experimental): Patients will receive three follow-up visits during the vulnerable period (three month after hospital discharge) in the HF network (either cardiologist in private practice or HF outpatient clinic)
  Interventions: Other: Heart Failure network care
- Randomised Arm 2: Usual care (No Intervention): Patients will receive usual care by their primary physician or cardiologist
- Registry Arm for non-randomised patients (No Intervention): Patients not willing to be randomised will be followed in a registry.

INTERVENTIONS:
Other: Heart Failure network care — Patients will receive three visits within the first three months after randomization for improving heart failure therapy at a cardiologist or the outpatient heart failure clinic
  Arms: Randomised Arm 1: Heart Failure Network Care

SUMMARY:
PEDAL-HF is a registry-based randomized prospective multicenter study. We plan to include 1000 patients who were recently admitted with acute decompensated heart failure at five tertiary heart clinics in Germany. For the randomised part, 750 patients will be randomized to care within a heart failure network or usual care. The primary endpoint of the randomized trial is change in NT-proBNP from baseline to 6 months of follow-up.

All patients (randomized or not) will be followed for two years.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the participating study centres with acute decompensated heart failure (ADHF), defined as clinical signs and/or symptoms of heart failure, objective structural cardiac abnormalitites according to the ESC criteria.

Exclusion Criteria:

* Age < 18 years, pregnancy, any condition interfering with the informed consent process, patients placed in an institution by official or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP plasma levels between baseline and 6 months visit | 6 months
  Adjusted geometric mean ratio between 6 months visit and baseline visit

SECONDARY OUTCOMES:
Change in KCCQ from baseline to 6 months of Follow-up | 6 months
  Quality of life measured by Kansas City Cardiomyopathy Questionnaire

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared following reasonable scientific request